CLINICAL TRIAL: NCT02622139
Title: Monocentric, Prospective Interventional Study to Assess the Degree of Disease Activity With a Multispectral Optoacoustic Tomography (MSOT) Handheld Scanner in Patients With Crohn's Disease or Ulcerative Colitis
Brief Title: Multispectral Optoacoustic Tomography (MSOT) for the Evaluation of Disease Activity in Inflammatory Bowel Diseases (IBD)
Acronym: MSOT_IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: iThera Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 252_15B
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis; IBD
Keywords: Photoacoustics; Optoacoustics; Ultrasound
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multispectral Optoacoustic Tomography (Experimental): Multispectral Optoacoustic Tomography (MSOT) for the evaluation of disease activity in inflammatory bowel diseases (IBD)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — MSOT for the evaluation of disease activity in IBD patients

SUMMARY:
Monocentric, prospective interventional study to assess the degree of disease activity with a multispectral optoacoustic tomography (MSOT) handheld scanner in patients with Crohn's disease or ulcerative colitis.

DETAILED DESCRIPTION:
The proposed study is designed as a pilot study to evaluate the usefulness of MSOT for the evaluation of disease activity in IBD patients. As current methods for the evaluation of intestinal inflammation in IBD have relevant restrictions, new, non-invasive, quantitative, and accurate modalities are urgently needed. In comparison to other techniques, MSOT provides relevant advantages such as non-invasive imaging, high spatial resolution (this is of special importance for the evaluation of the intestine, which can be only a few millimeters thick), and highly sensitive detection of specific molecules such as total hemoglobin or oxy- /deoxygenated hemoglobin. These advantages suggest MSOT as an outstanding technique for evaluating disease activity in IBD.

The proposed study incorporates nearly no risk for participating patients and might provide relevant data for more a more in depth analysis of MSOT for IBD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Histological verified Crohn's disease or ulcerative colitis
* Age > 18 years

Exclusion Criteria:

* Age < 18 years
* Mental retardation of the patient with restriction of general judgment and awareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Correlation of MSOT-data with clinical activity scores of IBD | 12 month
Correlation of MSOT-data with sonographic parameters | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Department 1, University of Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knieling F, Neufert C, Hartmann A, Claussen J, Urich A, Egger C, Vetter M, Fischer S, Pfeifer L, Hagel A, Kielisch C, Gortz RS, Wildner D, Engel M, Rother J, Uter W, Siebler J, Atreya R, Rascher W, Strobel D, Neurath MF, Waldner MJ. Multispectral Optoacoustic Tomography for Assessment of Crohn's Disease Activity. N Engl J Med. 2017 Mar 30;376(13):1292-1294. doi: 10.1056/NEJMc1612455. No abstract available. PMID 28355498
- [Result] Waldner MJ, Knieling F, Egger C, Morscher S, Claussen J, Vetter M, Kielisch C, Fischer S, Pfeifer L, Hagel A, Goertz RS, Wildner D, Atreya R, Strobel D, Neurath MF. Multispectral Optoacoustic Tomography in Crohn's Disease: Noninvasive Imaging of Disease Activity. Gastroenterology. 2016 Aug;151(2):238-40. doi: 10.1053/j.gastro.2016.05.047. Epub 2016 Jun 3. No abstract available. PMID 27269244